CLINICAL TRIAL: NCT02731443
Title: The Impact of Epilepsy Surgery on Dream Content
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, David Steven, David A. Steven, MD, MPH, FRCSC, FACS, London Health Sciences Centre
Other Study IDs: 107654
Record Dates: First submitted 2016-04-02; First posted 2016-04-07 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Dream Content
Keywords: dreaming; epilepsy; neurosurgery; temporal lobectomy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ESx: Epilepsy patients undergoing elective surgical resection of brain tissue; study group: epilepsy surgery=ESx.
  Interventions: Procedure: Epilepsy surgery
- DE: Epilepsy patients undergoing elective depth electrodes insertion in general anesthesia; control group: depth electrodes=DE.
  Interventions: Procedure: Depth electrodes insertion

INTERVENTIONS:
Procedure: Epilepsy surgery — Epilepsy surgery is a procedure that removes an area of the brain where seizures originate.
  Groups: ESx
Procedure: Depth electrodes insertion — Depth electrodes are inserted for monitoring/mapping the subsurface levels of the brain for the surgical treatment of epilepsy.
  Groups: DE

SUMMARY:
Prospective observational study on epilepsy patients undergoing partial brain resection surgery (i.e. anterior temporal lobectomy) to assess the change in dream content before and 3 months and 1 year after surgery using anonymized dream-recall questionnaires. A control group of epilepsy patients undergoing diagnostic depth electrodes placement will complete the same questionnaires pre- and postoperatively to asses the factor 'general anesthesia' as a potential confounder.

DETAILED DESCRIPTION:
STUDY RATIONALE Dream research, unlike sleep research, has not greatly developed anymore as there are few dream research laboratories only and not much systematic dream research is done outside the laboratory either(1) although validated methods of collecting and analyzing dream reports on the basis of the coding system developed by Calvin S. Hall and Robert Van de Castle are readily available.(2) According to Domhoff et al.,(3) the main features of the default dream network include the medial prefrontal cortex, the medial temporal lobe, the bilateral inferior parietal lobule/temporoparietal junction, and the posterior cingulate cortex, with the medial pre- frontal cortex and the posterior cingulate cortex serving as major hubs. The dorsal medial subsystem including the dorsomedial prefrontal cortex, the temporoparietal junction/anterior inferior parietal lobule, the lateral temporal cortex, and temporopolar cortex (the anterior pole of the temporal lobe) is activated by instructions to think about the present situation or a present mental state (''present self'').(3) The medial temporal subsystem including the ventral medial prefrontal cortex, posterior inferior parietal lobule, retrosplenial cortex, parahippocampal cortex, and hippocampal formation is activated by thinking about personal situations and decisions in the future (''future self'').(3) A lot of what is known about the neuronal function of dreaming comes from lesion studies that are well-summarized by Solms.(4) To the best knowledge, investigators are the first to prospectively investigate the change of dream content in patients electively undergoing surgical resection of brain tissue (i.e. the anterior temporal lobe for temporal lobe epilepsy).

The merits of the current study are the following:

* To better understand the dream network (academic significance)
* To better consult epilepsy patients with respect to the impact of surgery on dreaming (practical significance)

PURPOSES AND OBJECTIVES

Purpose:

- To assess the change in dream content in patients following epilepsy surgery compared to a control group of patients undergoing general anesthesia.

Hypothesis:

- Dream content is markedly changed in patients before and after epilepsy surgery.

Objective:

- To quantify dream content in patients before and after epilepsy surgery using the MOST RECENT DREAM questionnaire and compare these results to patients undergoing general anesthesia (control group).

STUDY DESIGN AND METHODOLOGY Setting/Design: Prospective observational study on epilepsy patients undergoing elective surgical resection of brain tissue (study group: Epilepsy surgery=ESx) or depth electrode insertion in general anesthesia (control group=DE).

Methodology: Patient baseline characteristics are Age (minimum age: 16 years); Date of birth (DOB); Sex; Handedness: RH/LH; Education (years); Occupation according to the International Standard Classification of Occupation(5); Seizure history (years); Seizure frequency ENGEL classification; Antiepileptic drugs; Other medication (antidepressants, dopaminergic agonists and antagonists, etc.); Pathology (Ammon's horn sclerosis y/n); Side (right/left); Any previous cranial surgery; Other relevant medical history (dementia, depression and other psychiatric disorders, Parkinson's, etc.) Questionnaire: MOST RECENT DREAM (STANDARD INSTRUMENT (2)

STUDY PROCEDURES AND SPECIFIC TESTINGS In this observational study, the MOST RECENT DREAM questionnaire, a standard validated instrument(2) represents the only study specific testing outside of standard care. The questionnaire is handed out to patients to record the most recent dreams five times pre- and post-operatively. The length of each dream summary lies in between 50 and 300 words. Study participation and the questionnaires will not affect standard patient care in any way and carries no additional risks.

STUDY GROUP:

Visit 1 (pre-op outpatient clinics or epilepsy monitoring unit) - Study information - Informed consent - Hand-out anonymized MOST RECENT DREAM (5x), return by mail before surgery.

Visit 2 (post-op outpatient clinics at ~1 month) - Hand-out anonymized MOST RECENT DREAM (5x) to be completed and returned by mail at 3 months postoperatively - Outcome according to the Engel classification Long-term FU at 12 month - Mail anonymized MOST RECENT DREAM (5x), return by mail.

CONTROL GROUP (Diagnostic depth electrodes):

Visit 1 (pre-op outpatient clinics/epilepsy monitoring unit) Study information - Informed consent - Hand-out anonymized MOST RECENT DREAM (5x), return before surgery.

Visit 2 (post-op epilepsy monitoring unit) Hand-out anonymized MOST RECENT DREAM (5x) to be completed and returned by mail at 1 month postoperatively.

DATA ANALYSIS Major indicators for main content categories in the Hall/Van de Castle system(2) are compared before and after the index procedure and results will be presented graphically similar to Bentes et al.(6). Data analysis is done using EXCEL spreadsheets available from http://www.dreamresearch.net/ and analysis performed as explained at http://www2.ucsc.edu/dreams/Info/statistics.html

ELIGIBILITY:
Inclusion Criteria:

* All epilepsy patients (minimum age: 16 years) undergoing elective surgical resection of brain tissue (study group) or depth electrode insertion in general anesthesia (control group) that give written consent after thorough study information.
* Patients must be able to understand the study concept and willing/able to document their most recent dream in written.

Exclusion Criteria:

* Inability to document their most recent dream in written (language barrier, illiteracy, low intelligence, mental disabilities). Age <16 years.
* Relevant co-morbidities such as dementia, depression and other psychiatric disorders, Parkinson's disease.
* Previous cranial surgery in a relevant cortical area of the default dream network.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Epilepsy patients undergoing elective surgical resection of brain tissue (study group: Epilepsy surgery=ESx) or depth electrode insertion in general anesthesia (control group=DE).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage Change of Dream Features Occurrence (i.e. dream content; MOST RECENT DREAM questionnaire) - both groups (ESx & control group) | 3 months
  Percentage change of the following dream features occurrences according to the Hall/Van de Castle system are considered:
  * Characters
  * Social Interactions
  * Aggression
  * Friendliness
  * Sexuality
  * Activities (walking, talking, seeing, thinking, etc.)
  * Success and Failure
  * Misfortune and Good Fortune
  * Emotions
  * Settings
  * Objects
  * Descriptive Elements (modifiers, time, negatives)
  The relative abundance of the dream content listed above will be expressed in percentage and postoperative changes compared to the preoperative baseline.
  Relative differences between the indicators will be determined and statistically tested for significance. The one indicator that turns out to be statistically different from the rest will be considered the primary outcome measure. For an example, compare Bentes et al. 2011.

SECONDARY OUTCOMES:
Dream Content (MOST RECENT DREAM questionnaire) - ESx group | 12 months
  Major indicators for main content categories according to the Hall/Van de Castle system.

OTHER OUTCOMES:
Seizure frequency (ESx only) | 3 and 12 months
  According to the ENGEL classification
Anti epileptic drugs (AED) usage (ESx only) | 3 and 12 months
  Number of different AED

CONTACTS AND LOCATIONS:
Overall Officials: David A Steven, M.D., Principal Investigator — London Health Science Center
Locations (1):
- London Health Sciences Center, University Hospital, London, Ontario, Canada

REFERENCES:
- [Result] Domhoff GW, Schneider A. New rationales and methods for quantitative dream research outside the laboratory. Sleep. 1998 Jun 15;21(4):398-404. doi: 10.1093/sleep/21.4.398. PMID 9646385
- [Result] Schneider A, Domhoff GW. The Quantitative Study of Dreams. Retrieved December 13 2015: http://www.dreamresearch.net/.
- [Result] Domhoff GW, Fox KC. Dreaming and the default network: A review, synthesis, and counterintuitive research proposal. Conscious Cogn. 2015 May;33:342-53. doi: 10.1016/j.concog.2015.01.019. Epub 2015 Feb 24. PMID 25723600
- [Result] Solms M. Dreaming and REM sleep are controlled by different brain mechanisms. Behav Brain Sci. 2000 Dec;23(6):843-50; discussion 904-1121. doi: 10.1017/s0140525x00003988. PMID 11515144
- [Result] International Standard Classification of Occupations (ISCO). http://www.ilo.org/public/english/bureau/stat/isco/. Accessed 1st of August 2015.
- [Result] Bentes C, Costa J, Peralta R, Pires J, Sousa P, Paiva T. Dream recall frequency and content in patients with temporal lobe epilepsy. Epilepsia. 2011 Nov;52(11):2022-7. doi: 10.1111/j.1528-1167.2011.03290.x. Epub 2011 Oct 17. PMID 22003885